CLINICAL TRIAL: NCT00687622
Title: An Open-Label, Multiple-Dose, Dose-Escalation Study to Investigate the Safety, Pharmacokinetics, and Pharmacodynamics of the MEK Inhibitor GSK1120212 in Subjects With Solid Tumors or Lymphoma
Brief Title: Open-label Study to Investigate the Safety, PK, and Pharmacodynamics of GSK1120212 in Subjects With Solid Tumors or Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEK111054
Record Dates: First submitted 2008-05-28; First posted 2008-06-02 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Solid Tumours
Keywords: MEK inhibitor; solid tumors; First Time in Human; GSK1120212; Oncology; melanoma
MeSH Terms: conditions — Neoplasms; Melanoma | interventions — trametinib

ARMS (1):
- GSK1120212 (Experimental): Part 1 will identify the maximum tolerated dose using a dose-escalation procedure. Part 2 will explore further the safety, tolerability, and clinical activity of GSK1120212 in subjects with pancreatic, melanoma, non-small cell lung, and KRAS or BRAF mutation-positive colorectal cancer. Part 3 will characterize the range of biologically effective doses by assessing pharmacodynamic markers in tumor tissue
  Interventions: Drug: GSK1120212

INTERVENTIONS:
Drug: GSK1120212 — Part 1-dose-escalation Part 2 - Recommended Part 2 dose Part 3 - characterize the range of biologically effective doses

SUMMARY:
MEK111054 is a first-time-in-human, open-label study to determine recommended dose and regimen for the orally administered GSK1120212. The study consists of three parts. Part 1 will identify the maximum tolerated dose. Part 2 will explore the safety, tolerability, and effectiveness of GSK1120212. Part 3 will determine a range of effective doses.

ELIGIBILITY:
Inclusion Criteria:

Part 1

* Written informed consent provided.
* 18 years old or older.
* Histologically or cytologically confirmed diagnosis of solid tumor malignancy or lymphoma that is not responsive to standard therapies or for which there is no approved or curative therapy.
* Performance Status score of 0 or 1 according to the Eastern Cooperative Oncology Group (ECOG) scale.
* Able to swallow and retain oral medication.
* Male subjects must agree to use one of the contraception methods listed. This criterion must be followed from the time of the first dose of study medication until four weeks after the last dose of study medication. However, the Sponsor advises that contraception be used for a total of 16 weeks following the last dose (based on the lifecycle of sperm).
* A female subject is eligible to participate if she is of:

  * Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/mL and estradiol < 40 pg/mL (<140 pmol/L) is confirmatory]. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods in Section 8.1 if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least two to four weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.
  * Child-bearing potential and agrees to use one of the contraception methods listed in Section 8.1 for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until four weeks after the last dose of study medication.
  * Note: Oral contraceptives are not reliable due to potential drug-drug interaction.
* CPP</= 4.0 mmol2/L2 (55 mg2/dL2)
* Adequate organ system function as defined in Table 9. Absolute neutrophil count (ANC)>/= 1.0 X 109/L; Hemoglobin >/= 9 g/dL; Platelets >/= 75 X 109/L; PT/INR and PTT </= 1.3 X ULN; Total bilirubin </=1.5 mg/dL; AST and ALT </= 2.5 X ULN (can be higher in the presence of liver metastasis.); Creatinine </= ULN OR Calculated creatinine clearance >/= 50 mL/min OR 24-hour urine creatinine clearance >/= 50 mL/min; Ejection fraction >/= LLN by ECHO or MUGA.

Part 2 - As per Part 1 with the exception of criterion 3 and:

* Histologically or cytologically confirmed diagnosis of melanoma, pancreatic, colorectal cancer (CRC), non-small cell lung cancer, or other tumor with BRAF mutation.
* CRC must be KRAS or BRAF mutation positive.
* Subjects with melanoma, CRC, or non-small cell lung cancer must provide either the results of a BRAF or KRAS mutation assay, archived tumor tissue, or a fresh biopsy.
* Subjects must be incurable or resistant to standard therapy.

Part 3 - As per Part 1 and:

* For the biopsy portion of the study, subjects must have accessible tumor for biopsy, and willingness to provide pre- and post dose biopsies.

Exclusion Criteria:

* Currently receiving cancer therapy (chemotherapy, radiation therapy, immuno-therapy, biologic therapy, hormonal therapy, surgery and/or tumor embolization).
* Use of an investigational anti-cancer drug within 28 days or five half-lives, whichever is shorter, prior to the first dose of GSK1120212. A minimum of 10 days between termination of the investigational drug and administration of GSK1120212 is required. In addition, any drug-related toxicity should have recovered to Grade 1 or less.
* Previous treatment with a MEK inhibitor. Subjects previously treated with a BRAF inhibitor are eligible with approval of a GSK medical monitor.
* Current use of a prohibited medication or requires any of these medications during treatment with GSK1120212.
* Current use of warfarin. NOTE: Low molecular weight heparin and prophylactic low-dose warfarin are permitted. PT/PTT must meet the inclusion criteria. Subjects taking warfarin must have their INR followed closely.
* Presence of active gastrointestinal disease or other condition that will interfere significantly with the absorption, distribution, metabolism, or excretion of drugs.
* Any major surgery, radiotherapy, or immunotherapy within the last four weeks. Chemotherapy regimens with delayed toxicity within the last four weeks (six weeks for prior nitrosourea or mitomycin C). Chemotherapy regimens given continuously or on a weekly basis with limited potential for delayed toxicity within the last two weeks. Note: Use of erythropoietin replacement or bisphosphonates is considered supportive care and their use is permitted.
* History of RVO or central serous retinopathy.
* Visible retinal pathology as assessed by ophthalmologic exam that is considered a risk factor for retinal vein thrombosis or central serous retinopathy.
* Intraocular pressure > 21mm Hg as measured by tonography.
* Glaucoma diagnosed within one month prior to study Day 1.
* Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol.
* Concurrent condition that in the investigator's opinion would jeopardize compliance with the protocol.
* Leptomeningeal metastases or spinal cord compression due to disease.
* Subjects with previously untreated brain metastases. Subjects with brain metastases that were previously treated with gamma knife or whole brain radiation may enroll two weeks or four weeks after treatment, respectively. These subjects must be asymptomatic and either off corticosteroids or on a stable dose of corticosteroids for at least one month prior to the first dose of GSK1120212. Subjects are not permitted to receive enzyme inducing anti-epileptic drugs (EIAEDs) during the study.
* Primary malignancy of the central nervous system.
* Evidence of severe or uncontrolled systemic diseases (e.g., unstable or uncompensated respiratory, hepatic, renal, or cardiac disease).
* Unresolved toxicity greater than common terminology criteria for adverse events (CTCAE) Grade 1 from previous anti-cancer therapy except alopecia (if applicable) unless agreed to by a GSK Medical Monitor and the investigator.
* QTc interval >/= 480 msecs.
* History of acute coronary syndromes (including unstable angina), coronary angioplasty, or stenting within the past 24 weeks.
* Class II, III, or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system.
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to the study drug, dimethyl sulfoxide (DMSO), or excipients.
* Pregnant or lactating female.
* Unwillingness or inability to follow the procedures outlined in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2008-07-28 (Actual); Primary Completion 2011-06-07 (Actual); Study Completion 2011-11-08 (Actual)

PRIMARY OUTCOMES:
- To determine the maximum tolerated dose of GSK1120212 | at each visit, throughout Part 1

SECONDARY OUTCOMES:
- To characterize the PK of GSK1120212 after single and repeat-dose administration | at each cycle, throughout the study
- To evaluate the pharmacodynamic response in tumors after treatment with GSK1120212 | screening and Cycle 1 Day 15 in Parts 1 and 3
- To explore relationships between GSK1120212 PK, MAPK signalling inhibition and clinical endpoints | screening and Cycle 1 Day 15
- To explore the clinical tumor response after treatment with GSK1120212 | throughout the study
- To determine the association of clinical and PK endpoints with genetic and protein profiles from tumor tissue | throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (12):
- United States (12):
  - GSK Investigational Site, Scottsdale, Arizona
  - GSK Investigational Site, Aurora, Colorado
  - GSK Investigational Site, Fort Myers, Florida
  - GSK Investigational Site, Ocoee, Florida
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Albany, New York
  - GSK Investigational Site, Kettering, Ohio
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Norfolk, Virginia

REFERENCES:
- [Background] Falchook GS, Lewis KD, Infante JR, Gordon MS, Vogelzang NJ, DeMarini DJ, Sun P, Moy C, Szabo SA, Roadcap LT, Peddareddigari VG, Lebowitz PF, Le NT, Burris HA 3rd, Messersmith WA, O'Dwyer PJ, Kim KB, Flaherty K, Bendell JC, Gonzalez R, Kurzrock R, Fecher LA. Activity of the oral MEK inhibitor trametinib in patients with advanced melanoma: a phase 1 dose-escalation trial. Lancet Oncol. 2012 Aug;13(8):782-9. doi: 10.1016/S1470-2045(12)70269-3. Epub 2012 Jul 16. PMID 22805292
- [Background] Infante JR, Fecher LA, Falchook GS, Nallapareddy S, Gordon MS, Becerra C, DeMarini DJ, Cox DS, Xu Y, Morris SR, Peddareddigari VG, Le NT, Hart L, Bendell JC, Eckhardt G, Kurzrock R, Flaherty K, Burris HA 3rd, Messersmith WA. Safety, pharmacokinetic, pharmacodynamic, and efficacy data for the oral MEK inhibitor trametinib: a phase 1 dose-escalation trial. Lancet Oncol. 2012 Aug;13(8):773-81. doi: 10.1016/S1470-2045(12)70270-X. Epub 2012 Jul 16. PMID 22805291
- See also: Results for study MEK111054 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/MEK111054?search=study&study_ids=MEK111054#rs